CLINICAL TRIAL: NCT05152446
Title: Implementation of an Infusion Management Scheme to Improve Patient Outcome in Tertiary Children's Hospitals：A Multi-center Before-afer Trial
Brief Title: Implementation of an Infusion Management Scheme to Improve Patient Outcome in Tertiary Children's Hospitals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital (Other); Anhui Provincial Children's Hospital (Other); Dalian women and children's medical group (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); Qidong Women's and Children's Health (Unknown); Chengdu Women's and Children's Central Hospital (Other); Hunan Children's Hospital (Other Government); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FNDGJ202110
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Children,Hospitalized; Infusion; Infections
Keywords: implementation study; pediatric; effect evaluation; management of infusion nursing
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infusion management scheme (Experimental): To implement infusion management scheme, then observe the continuous changes.
  Interventions: Other: Infusion management scheme

INTERVENTIONS:
Other: Infusion management scheme — * To set up a pediatric intravenous infusion team;
  * To form standardized procedures by carrying out a quality improvement program in collecting and sending samples for inspection once suspected CLABSI occurs (1 month for training and 3 months for continuous improvement ); providing infusion training curriculums to nurses in forms of lectures, group discussions, operation demonstrations, and scenario simulations, holding practice review meeting with them; providing elements to caregivers of educational leaflet, nurse-provided education during patients' infusion therapy( 6-month implementation);
  * To observe the continued daily infusion practice in 6 months.

SUMMARY:
This study is a multi-center before-after trial design. The object is to observe whether the incidence of central line associated blood stream infection(CLABSI) will tend to descend compared with retrospective electronic medical record data after implementation of an infusion management scheme which comes form " Clinical Practice Guideline on Infusion Therapy in Children " .

DETAILED DESCRIPTION:
Infusion therapy is an important part in pediatric ward. Most hospitalized children need indwelling vascular access devices to receive infusion therapy. Much attention has been paid to possible serious or fatal complications due to immature immune system, poor communication ability and cognitive disorder in children during catheter placement, use and maintenance. Reducing the complications related to central venous catheter has become the focus of the global health care system. Studies have shown that the technical level of operators is in connection with the incidence of CLABSI, and an intravenous infusion team (IV Team) is the key to preventing CLABSI, which may fundamentally improve the clinical outcomes of pediatric patients. From December 2021 to April 2023, taking Children's Hospital of Fudan University as the leading center, Xiamen Children's Hospital, Anhui Provincial Children's Hospital, Dalian Municipal Women and Children's Medical Group, Tongji Hospital, First Affiliated Hospital of Guangxi Medical University, Qidong Women's and Children's Health, Chengdu Women's and Children's Central Hospital, Hunan Children's Hospital as the cooperation centers. A retrospective review of electronic medical record data will be collected first. The intervention is composed of setting up a pediatric intravenous infusion team; carrying out a quality improvement in collecting and sending suspected CLABSI samples; providing infusion training curriculums to nurses in forms of lectures, group discussions, operation demonstrations, and scenario simulations, holding practice review meeting with them; providing elements to caregivers of educational leaflet, nurse-provided education during patients' infusion therapy.

ELIGIBILITY:
Inclusion Criteria for centers:

* A tertiary children's hospital with more than 300 beds
* The vice president in charge of nursing affairs, the director of nursing department and the director of hospital infection control department all agree in participating in this study with written permission, which include total acceptance of infusion management scheme and outcome indicators report as required
* To obtain the approval from Ethics Committee of the hospital

Inclusion Criteria for patients:

* Hospitalized children aged 0~18 years
* Catheterization and maintenance in the same center
* The indwelling time is longer than 48h

Exclusion Criteria:

* The vice president in charge of nursing affairs or the director of nursing department inform the researcher to withdraw from this study with written form and should clear reasons
* The number of cases for suspected CLABSI sample actually submitted for inspection / The number of cases for suspected CLABSI sample should submitted for inspection<0.9
* The awareness rate of infusion management scheme in clinical nurses is less than 90% and the qualification rate of the practice examination in clinical nurses is less than90% during inspection

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of CLABSI | During the 6-month implementation
  CLABSI diagnostic criteria requires that a central line is in situ at the time of or within 48 hours; children with a central line have fever (over 38℃), chills, hypotension or mental state changes; there is no alternate source of bloodstream infection. Apart from the above three necessary requirements, CLABSI diagnosis could be accompanied by two positive blood cultures drawn from a peripheral vein and a CVAD, two positive blood cultures drawn from different CVADs, one positive blood culture from a CVAD with a planned specific antimicrobial therapy or common skin contamination bacteria cultured (eg. Coagulase-negative Staphylococci, diphtheroids, Bacillus or Micrococcus).
  Incidence of CLABSI = (case numbers of CLABSI)/(Catheter Days per Month)×1000‰.

SECONDARY OUTCOMES:
Changes of Inspection rate of suspected CLABSI samples | From baseline to the end of the 6-month implementation
  When there are suspected cases of CLABSI, the physician will prescribe blood culture and the nurse will draw blood within 1 hour and send them for inspection (if antibiotics are needed, blood should be drawn before administration).
  Suspected CLABSI samples inspection rate= (documented samples for inspection )/(Required samples for inspection)×100%.
Incidece of infiltration (of Grade2 or higher) and/or extravasation | During the 6-month implementation
  Incidence of infiltration (of Grade2 or higher) and extravasation: The bedside nurses document PIV infiltration and extravasation using "Pediatric PIV Infiltration Scale" during fluid infusing and every shift.
  Incidence of infiltration (of Grade2 or higher) and/or extravasation = (case numbers of infiltration (of Grade2 or higher) and/or extravasation)/(Catheter Days per Month)×1000‰.
Changes of the scores of readiness of internal context | From baseline to the end of the 6-month implementation
  10% of nurses in every participant center will be randomly drawn to complete the investigation questionnaire for the readiness of internal context using self-made "Assessment Tool of Organizational Internal Context (6 items) " and "Assessment Tool of Local Internal Context ( 9 items)".The purpose of the survey is to evaluate the internal context of evidence-based practice in each participant center. The score of each item is based on Likert 5 grades rating levels from 1 (lowest) to 5 (highest).

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Xiamen Children's Hospital, Xiamen, Fujian
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Qidong Women's and Children's Health, Qidong, Jiangsu
  - Dalian women and children's medical group, Dalian, Liaoning
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No